CLINICAL TRIAL: NCT00623090
Title: Internet-Based Education for Prostate Cancer Screening
Acronym: PCSEd
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kathryn L. Taylor, Ph.D., Associate Professor, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: PC051100; R01CA119168-01 (NIH)
Record Dates: First submitted 2008-02-14; First posted 2008-02-25 (Estimated); Last update posted 2012-12-13 (Estimated); Status verified 2012-12

CONDITIONS: Prostate Cancer
Keywords: prostate cancer screening education; behavioral oncology; randomized trial
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 Website (Experimental): Participants receive the Login information for the Internet we developed on prostate cancer screening.
  Interventions: Behavioral: educational internet site on prostate cancer screening
- 2 Booklet (Active Comparator): Participants receive the education booklet we developed on prostate cancer screening.
  Interventions: Behavioral: Educational print booklet
- 3 Usual Care (Placebo Comparator): Usual care: participants receive no intervention.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: educational internet site on prostate cancer screening — Healthy men between 45-70 receive the login information to access our educational internet site on prostate cancer screening.
  Arms: 1 Website
Behavioral: Educational print booklet — Healthy men between 45-70 receive a copy of our educational print booklet in the mail.
  Arms: 2 Booklet
Behavioral: Usual care — Healthy men aged 45-70 receive no intervention and are followed for one year, along with the men in the two intervention arms.
  Arms: 3 Usual Care

SUMMARY:
Prostate cancer (PCa) is the leading cancer diagnosis among men and the second leading cause of male cancer death. However, screening asymptomatic men remains controversial, as early diagnosis and treatment of PCa has not yet demonstrated reduced disease-related mortality in a randomized trial. The goal of the current study is to develop and assess widely accessible methods to assist men in making informed decisions about PCa screening. We will compare the efficacy of a new web-based, interactive decision support approach to our existing print-based PCa screening decision tool, among a diverse sample of male primary care patients. Abundant evidence documents the expanding role of the Internet in increasing access to and understanding of health information and the need for systematic evaluations of Internet-based interventions. A novel aspect of the proposed trial will be our focus on cognitive biases as a factor that has limited the success of previous information-based interventions. Specifically, we will evaluate: 1) confirmation bias and 2) short-term consequences bias.

DETAILED DESCRIPTION:
In Phase I (months 1-8) of this five-year project, we will develop an interactive, Internet-based, patient information and decision aid. In Phase II (months 9-60), we will evaluate the impact of this decision aid in a randomized controlled trial with male primary care patients aged 45-70 from three Washington, District of Columbia area health care settings (N = 1875). Trial arms include: 1) print-based information and decision aid (Print), 2) web-based information plus interactive decision aid (Web), and 3) usual care (UC). Subjects will complete outcome assessments at baseline, one- and 13-months post-baseline. The specific aims are to: 1. Evaluate the impact of the delivery method (Web vs. Print vs. Usual Care) on the key patient outcome variables of knowledge, decisional satisfaction, and the screening decision. 2. Identify factors that moderate the interventions' impact on the primary outcomes. 3. Identify the mechanisms by which the interventions impact knowledge and decisional satisfaction. In exploratory analyses, we will evaluate factors that are related to use of the web and print materials. This research has the potential to make several significant and innovative contributions: 1) the development and evaluation of a widely accessible method of educating a heterogeneous group of patients about a controversial topic, which can be adapted for other similarly contentious issues, 2) a determination of whether Web based materials are a feasible method of patient education for this age cohort, compared to print materials, 3) an understanding of cognitive factors that may hinder comprehension of a controversial medical decision, 4) a determination of who among the target population benefits the most from a web-based intervention, and 5) the information required to streamline and target future web-based educational interventions.

ELIGIBILITY:
Inclusion Criteria:

* Active primary care patients at Georgetown University Medical Center, Washington Hospital Center, or Medstar Physician Partners (I,e, seen during the past two years)
* English-speaking
* 45-70 years of age; AND
* Ability to provide meaningful consent.

Exclusion Criteria:

* History of prostate cancer.

Ages: 45 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1893 (Actual)
Dates: Start 2007-10; Primary Completion 2011-03 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
screening decision | one-year follow up
knowledge about prostate cancer screening | one-month and one-year post-intervention
decisional satisfaction | one-month and one-year post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn L. Taylor, PhD, Principal Investigator — Georgetown University
Locations (2):
- United States (2):
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Washington Hospital Center, Washington D.C., District of Columbia

REFERENCES:
- [Derived] Dorfman CS, Williams RM, Kassan EC, Red SN, Dawson DL, Tuong W, Parker ER, Ohene-Frempong J, Davis KM, Krist AH, Woolf SH, Schwartz MD, Fishman MB, Cole C, Taylor KL. The development of a web- and a print-based decision aid for prostate cancer screening. BMC Med Inform Decis Mak. 2010 Mar 3;10:12. doi: 10.1186/1472-6947-10-12. PMID 20199680